CLINICAL TRIAL: NCT04623983
Title: 3D Printed Indirect Bonding Trays - Accuracy of Rigid Versus Resilient Resin a Clinical in Vivo Study
Brief Title: Accuracy of 3D Printed Indirect Bonding Trays - an in Vivo Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Nemec, Staff member, dentist, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1485/2020
Record Dates: First submitted 2020-10-08; First posted 2020-11-10 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Dental Bonding

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- resilient bonding tray (Experimental): Patients receiving resilient orthodontic bonding trays
  Interventions: Device: bonding tray
- rigid bonding tray (Experimental): Patients receiving rigid orthodontic bonding trays
  Interventions: Device: bonding tray

INTERVENTIONS:
Device: bonding tray — Orthodontic bonding tray
  Other Names: Ortho Rigid Bonding tray

SUMMARY:
Objective In addition to examining the transmission accuracy of rigid and non-rigid IDB's the aim of the study is to determine the 'lost rate' during the placement. The 'lost rate' is the percentage frequency of brackets that have no adhesion to the model after the bonding has taken place.

Hypothesis The main hypothesis does not describe a significant deviation of the digitally planned to the actually placed bracket position in directions and angles described.

The secondary hypothesis is the assumption of no significant difference between the accuracy and lost rate of the two materials.

Method 24 orthodontic patients treated with multibracket appliance will be included for the planned study. In order to increase the reproducibility of the acquired data four different model situations are included.

Objective The aim of the study is a scientific examination of the accuracy of digital printed bonding trays using two materials to support the decision process of the potential user and their dental laboratories. The study allows an insight into the technical manufacturing process and its workflow.

DETAILED DESCRIPTION:
Orthodontic clinicians distinguish between direct and indirect brackets placement. Using the direct procedure, brackets are placed on the patients tooth without a transfer appliance. While the indirect method takes advantage of placing the brackets on a dental model under laboratory surrounding.

The conventional method of indirect bracket positioning uses plaster models from the treated dental arches. Following the positioned brackets are transferred from the model to the patient mouth using a so called indirect bonding trays (IDB). IDB's represent a transfer aid for the bracket placement. Advantages of this procedure can be an improvement of the tooth axis (facial axis) assessment especially since the model is freely movable in space further an optimized visibility with laboratory lighting. The placement on the digital model offers a variety of options with regards to measurement, magnification, contrast adjustment and exact referencing on the neighboring tooth.

Digital Workflow:

Under the broad term of rapid prototyping developments of applications allow a fully digital workflow while planning and manufacturing IDB's. The construction of bonding trays is based on a digital 3D model and is further manufactured using stereolithographic 3D printers. Similar to conventional IDB's there is the question of the optimal material with regards to transfer accuracy, dimensional stability and clinical applicability with 3D printed IDB's. Besides the question of transfer accuracy, the planned study will document the percentual number of brackets which failed to bond with the corresponding tooth (Lost Rate) using two different materials.

Objective:

The aim of the study is a scientific examination of the accuracy of digital printed bonding trays using two materials to support the decision process of the potential user and their dental laboratories. The study allows an insight into the technical manufacturing process and its workflow.

ELIGIBILITY:
Inclusion Criteria:

* Little Index 2,
* Little Index 3
* Little Index 4
* spacing

Exclusion Criteria:

* epilepsy
* periodontal disease
* infraocclusion
* agenesis
* tooth impaction

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy of indirectly placed brackets via indirect bonding trays | orthodontic bracket placement immediately after bonding
  3D Offset of indirectly bonded brackets

SECONDARY OUTCOMES:
Lost rate | orthodontic bracket placement immediately after bonding
  Non-bonded brackets

CONTACTS AND LOCATIONS:
Overall Officials: Erwin Jonke, MD, DMD, Study Chair — Medical University of Vienna; Alexander Schwaerzler, DMD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmid J, Brenner D, Recheis W, Hofer-Picout P, Brenner M, Crismani AG. Transfer accuracy of two indirect bonding techniques-an in vitro study with 3D scanned models. Eur J Orthod. 2018 Sep 28;40(5):549-555. doi: 10.1093/ejo/cjy006. PMID 29471483
- [Background] Castilla AE, Crowe JJ, Moses JR, Wang M, Ferracane JL, Covell DA Jr. Measurement and comparison of bracket transfer accuracy of five indirect bonding techniques. Angle Orthod. 2014 Jul;84(4):607-14. doi: 10.2319/070113-484.1. Epub 2014 Feb 20. PMID 24555689
- [Background] Oliveira NS, Gribel BF, Neves LS, Lages EMB, Macari S, Pretti H. Comparison of the accuracy of virtual and direct bonding of orthodontic accessories. Dental Press J Orthod. 2019 Sep 5;24(4):46-53. doi: 10.1590/2177-6709.24.4.046-053.oar. PMID 31508706
- [Derived] Schwarzler A, Nemec M, Lettner S, Rank C, Schedle A, Jonke E. 3D printed indirect bonding trays: Transfer accuracy of hard versus soft resin material in a prospective, randomized, single-blinded clinical study. Dent Mater. 2023 Nov;39(11):1058-1065. doi: 10.1016/j.dental.2023.09.011. Epub 2023 Oct 7. PMID 37806794